CLINICAL TRIAL: NCT05190991
Title: An International Multicenter Open-label Clinical Study of the Safety and Efficacy of RPH-104 for Prevention of Recurring Attacks in Adult Subjects With Familial Mediterranean Fever With Resistance to or Intolerance of Colchicine
Brief Title: Safety and Efficacy of RPH-104 Used to Prevent Recurrent Fever Attacks in Adult Patients With Colchicine Resistant or Colchicine Intolerant Familial Mediterranean Fever
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Atlant Clinical LLC (Unknown); Unimed Laboratories (Industry); Data Management 365 (Industry); R-Pharm JSC (Unknown); TRPharm İlaç Sanayi Ticaret Anonim Şirketi and ASCOT SCIENCE Education and Consulting Ltd. (Unknown); Exacte Labs LLC (Industry); Key Stat LLC (Unknown)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL04018071
Record Dates: First submitted 2021-11-03; First posted 2022-01-13 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Familial Mediterranean Fever; FMF
Keywords: RPH-104; colchicine inefficacy; colchicine intolerance; colchicine resistance; subcutaneous; FMF; interleukin-1 inhibitor
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RPH-104 q2w (Experimental): RPH-104 80 mg once every 2 weeks subcutaneously or RPH-104 160 mg once every 2 weeks subcutaneously
  Interventions: Biological: RPH-104

INTERVENTIONS:
Biological: RPH-104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial

SUMMARY:
The purpose of this study is to assess safety and efficacy of the long-term treatment with RPH-104 at doses of 80 or 160 mg once every 2 weeks (q2w) in patients with familial Mediterranean fever (FMF) with colchicine resistance or intolerance (i.e. colchicine resistant, crFMF), who completed the core study, during which they received at least one dose of RPH-104 (i.e. study patient population).

DETAILED DESCRIPTION:
This study is a long-term open-label extension (OLE) of the core double blind randomized placebo-controlled study CL04018065. This OLE study will have the following periods:

1. Screening period - 2 weeks (from signing an Informed Consent Form [ICF] at Visit 10 of the core study to Visit 1, Day 0 of this OLE study) - includes unblinding of the treatment groups determined in the core study (unless was unblinded previously) and determination of the eligibility criteria compliance for this study (all other screening procedures are performed after the completion of Visit 11 of the core study, which is also a Day 0 of this OLE study); All patients meeting the study inclusion/exclusion criteria according to the screening results will be transferred to the treatment period at the same day (Day 0) - the beginning of this period will be considered Visit 1 of this study
2. Treatment period - All patients will be receiving RPH-104 treatment for 198 weeks in the open-label regimen (both patient and the Investigator, along with all study team will know which treatment is used) at the doses determined for them in the core study. Thus, the possible RPH-104 dose will be:

   * 80 mg q2w subcutaneously (SC);
   * 160 mg q2w SC

   The first RPH-104 administration in this study will be performed at Visit 1. To maintain the q2w dosage regimen, the screening and the first open-label injection of RPH-104 (if the patient meets the study eligibility criteria) must be performed on the same day - Day 0 (which is also the day of Visit 11 of the core study) - i.e. the first administration in this study will be performed 2 weeks (±3 days) after the last administration in the core study.

   Further, RPH-104 will be administered to patients q2w both during each scheduled visit to the study site (with safety and efficacy assessments according to the visits schedule), and during Drug Administration Visits (DAVs) at the study site or at the patient's accommodation An injection of the study drug to patients is performed by qualified medical personnel every 2 weeks when the patient visits the study site; it is also possible for the patients to self-administer the drug at home (for which patients will be appropriately trained and provided with the necessary quantity of the drug, materials for the injection (including special containers for their disposal) and proper drug transportation).

   Safety and efficacy assessments are performed at Visit 1, Visit 2 (in 2 weeks), Visit 3 (in 4 weeks), Visit 4 (in 4 weeks), Visit 5 (in 8 weeks) and thereafter every 12 weeks (Visit 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20) according to the visits schedule. In case of RPH-104 administration in patients' accommodation, telephone contacts with a patient will be conducted by the Investigator every 4 weeks in between the visits starting from the Visit 4.In case of FMF attack development, patients who receive 80 mg of the drug may be switched to the increased maximum drug dose160 mg based at the discretion of the investigator.

   The drug is administered only at scheduled visits. Dose reduction of RPH-104 is not allowed in this study. After patients receive the last dose of RPH-104 at Week 198 of the study, the treatment period will be considered completed and an 8-week safety follow-up will start
3. Safety follow-up period - 8 weeks. During this period the patients will have to visit the study site twice in 4 weeks (Visit 21) and 8 weeks (Visit 22) after the last RPH-104 dose for safety assessments.

The last visit of the safety follow-up period (Visit 22) is the End of Study Visit; after completion of all procedures of this visit, patients will be considered to have completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient with Familial Mediterranean Fever (FMF) with resistance to or intolerance of colchicine, who completed the core study, during which he/she received at least one dose of RPH-104.
2. Voluntarily signed and dated Patient Informed Consent Form (ICF) for participation in this study.
3. The patient's ability and desire, according to the Investigator's discretion, to follow the schedule of visits, follow the study procedures and follow the Protocol requirements, including the following:

   * to visit the study site every 2 weeks for RPH-104 administration by qualified study site personnel

or

• to learn the subcutaneous (SC) injection technique and self-administer RPH-104 at his/her accommodation as per the study Protocol

or

• to agree with the qualified medical personnel visits to his/her accommodation for RPH-104 administration.

Exclusion Criteria:

1. Any medically significant event that was observed in a patient during his/her participation in the core study, as well as any other medical conditions (including psychiatric disorders) or laboratory abnormalities, which may increase the potential risk associated with participation in the study and treatment with RPH-104, or may affect the interpretation of the study results, and which, according to the Investigator's opinion, may lead to the patient's non-compliance with the study inclusion criteria.
2. Pregnant and/or lactating women or women planning pregnancy during the study or within 2 months after the last RPH-104 dose.
3. Women of childbearing potential, i.e. all females with physiological ability to conceive except for those with final cessation of menses, which should be determined retrospectively after 12 months of natural amenorrhea, i.e. amenorrhea with an appropriate clinical status, for example, at respective age, who do not agree to use highly effective contraceptives throughout the study, starting from the moment of signing the ICF and for at least 8 weeks after the last RPH-104 dose or Men who are sexually active and do not agree to use highly effective contraceptives throughout the study, starting from the moment of signing the ICF and for at least 8 weeks after the last RPH-104 dose.

   Highly effective contraception methods include:
   * complete abstinence: if it corresponds to the preferred and conventional lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation method) and interrupted coitus are not considered acceptable contraceptive methods;
   * female sterilization: surgical bilateral ovariectomy (with/without hysterectomy) or tubal ligation at least 6 weeks before the start of the core study. In a case of ovariectomy only, the female reproductive status should be verified by further hormonal test;
   * male sterilization (with documented absence of sperm in ejaculate post vasectomy) at least 6 months before the start of the core study. Vasectomized male partner should be the only partner of the participating female subject;
   * combination of any two of the following methods (a+b or a+c or b+c):

     1. use of oral, injectable or implanted hormonal contraceptives; in a case of oral contraceptives, the woman should constantly use the same product as was used during the core study;
     2. installation of an intrauterine device or contraceptive system;
     3. use of barrier contraceptives: condom or occlusive cap (diaphragm or cervical cap/contraceptive vaginal ring) with spermicidal foam/gel/film/cream/vaginal suppository
4. The need for a therapy with any of the following products from the moment of signing the ICF till the study treatment period completion:

   * systemic glucocorticoids at a dose exceeding 0,2 mg/kg/day of prednisolone (or 0,16 mg/kg/day of methylprednisolone, or an equivalent dose of another glucocorticoid) orally;
   * rilonacept, tocilizumab, rituximab, canakinumab, tumor necrosis factor alpha (TNF-a) inhibitors (TNFi) and other biological products (except for RPH-104);
   * immunosuppressants (cyclosporine, methotrexate, leflunomide, thalidomide, azathioprine, 6-mercaptopurine, cyclophosphamide, etc.);
   * methylprednisolone (or an equivalent) at a dose of more than 40 mg/day parenterally;
   * intramuscular, intra-articular or peri-articular administration of glucocorticoids;
   * anakinra;
   * tofacitinib, baricitinib;
   * any experimental drugs (except for RPH-104)
5. The need to use a live (attenuated) vaccine during the study or within 3 months after the last RPH-104 dose. Live attenuated vaccines include vaccines against viruses: measles, rubella, mumps, chickenpox, rotavirus, flu (as a nasal spray), yellow fever, polio (oral polio vaccine); vaccines against tuberculosis (BCG), typhoid fever (oral typhoid vaccine) and typhus (typhus vaccine). Immunocompetent family members of the patient should not be vaccinated with the oral polio vaccine during the patient's participation in the study
6. Positive results of tuberculosis screening performed at Visit 10 of the core study (QuantiFERON-Tuberculosis(TB)/T-Spot.TB test, chest X-ray).
7. Participation in other experimental studies (except for the core study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs), by System Organ Class and Preferred Term | Up to 62 weeks
Incidence of Treatment-Emergent Serious Adverse Events (SAEs), by System Organ Class and Preferred Term | Up to 62 weeks
Incidence of Treatment-Emergent Adverse Events of Special Interest (AESI), by System Organ Class and Preferred Term | Up to 62 weeks
Incidence rate for serious adverse events (SAEs) | Up to 62 weeks
  Incidence rate, expressed as the number of events per 100 patient-years of follow-up, for SAEs
Incidence rate for adverse events of special Interest (AESI) | Up to 62 weeks
  Incidence rate, expressed as the number of events per 100 patient-years of follow-up, for AESI

SECONDARY OUTCOMES:
Percentage of patients with physician global assessment of disease activity scale (PGA) <2 | Up to 62 weeks
  PGA of disease activity involves a 5-point system: from 0 = no clinical signs and symptoms associated with the disease to 4 = severe clinical signs and symptoms associated with the disease.
Percentage of patients with serological remission | Up to 62 weeks
  Serological remission is defined as C-reactive (CRP) level ≤10 mg/L.
Percentage of patients whose Serum amyloid A (SAA) levels returned to normal values | Up to 62 weeks
  SAA normal levels are defined as SAA <10 mg/L
Percentage of patients who have experienced ≥ 1 attacks per month (since Day 0) | Up to 54 weeks
  Criteria for the diagnosis of an attack are defined as the simultaneous development of clinical and serological signs of an attack, including:
  * the score on the scale of global physician's assessment of disease activity (PGA) ≥ 2, suggesting "mild", "moderate" or "severe" activity of the disease (i.e., clinical signs), AND
  * CRP level ≥ 30 mg/L (i.e. serological signs)
Percentage of patients who have not had a single attack | Up to 54 weeks
  Criteria for the diagnosis of an attack are defined as the simultaneous development of clinical and serological signs of an attack, including:
  * the score on the scale of global physician's assessment of disease activity (PGA) ≥ 2, suggesting "mild", "moderate" or "severe" activity of the disease (i.e., clinical signs), AND
  * CRP level ≥ 30 mg/L (i.e. serological signs)
Percentage of patients escalated to RPH-104 160 mg q2w dose | Up to 54 weeks
  The dose may be increased if a new attack is confirmed
Percentage of patients receiving additional symptomatic therapy with NSAIDs, paracetamol or glucocorticoids due to FMF | Up to 62 weeks
  Symptomatic therapy was prescribed by the decision of the investigator upon confirmation of a new attack
Change in the inflammatory markers CRP compared to baseline | Up to 62 weeks
  CRP level mg/l at each visit
Change in the inflammatory markers SAA compared to baseline | Up to 62 weeks
  SAA level mg/l at each visit
Changes in the PGA score over time | Up to 54 weeks
  PGA of disease activity involves a 5-point system: from 0 = no clinical signs and symptoms associated with the disease to 4 = severe clinical signs and symptoms associated with the disease.
Changes in the severity of chest pain based on the main disease symptoms scale. | Up to 54 weeks
  An assessment of severity of the main symptoms of the disease will be based on a 5-point scale: 0 = no symptom, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Changes in the severity of abdominal pain based on the main disease symptoms scale. | Up to 54 weeks
  An assessment of severity of the main symptoms of the disease will be based on a 5-point scale: 0 = no symptom, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Changes in the severity of arthralgia/arthritis based on the main disease symptoms scale. | Up to 54 weeks
  An assessment of severity of the main symptoms of the disease will be based on a 5-point scale: 0 = no symptom, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Changes in the severity of skin rash based on the main disease symptoms scale. | Up to 54 weeks
  An assessment of severity of the main symptoms of the disease will be based on a 5-point scale: 0 = no symptom, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Changes in the renal function in patients with impaired renal function at the screening | Up to 62 weeks
  Impaired renal function is defined as creatinine clearance(ClCr) <90 ml/min [calculated using the Cockcroft-Gault formula] at the screening
Changes in proteinuria in patients with baseline proteinuria | Up to 62 weeks
  Presence of protein in urine according to urinalysis results

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (8):
- Center of Medical Genetics and Primary Health Care LLC, Yerevan, Armenia
- Russia (4):
  - FSBEI HE First Moscow State Medical University named after I.M. Sechenov, Moscow
  - Moscow Multidisciplinary Scientific and Clinical Center named after S.P. Botkin, Moscow
  - Medical Technologies Ltd., Saint Petersburg
  - Terafarm, Llc, Stavropol
- Turkey (Türkiye) (3):
  - Hacettepe University Faculty of Medicine, Ankara
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul